CLINICAL TRIAL: NCT05739825
Title: Assessment Of Changes In Gut Microbiota Of Patients With Recurrent Clostridioides Difficile Infection After Fecal Microbiota Transplantation: Prospective Study
Brief Title: Changes in Recipients Gut Microbiota After Fecal Microbiota Transplantation
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, IANIRO GIANLUCA, Dr., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3555
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Clostridioides Difficile Infection Recurrence
Keywords: Clostridioides difficile infection; Fecal Microbiota Trasplantation; Engraftment
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — human feces. The human DNA will be discarded and not analysed at the time of the analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FMT from healthy donors — This intervention is represented by the administration, in the recipients' gut, of healthy donor microbiota through FMT

SUMMARY:
Clostridioides diﬃcile infection (CDI) is the most common cause of nosocomial diarrhea, and the most common health care-associated infectious disease in the United States, accounting for 15% of overall infections, nearly 30.000 deaths per year an estimated economic expense of $5 billion/year.

In the last decade, most of the burden related to CDI depends on recurrence CDI (rCDI) (3). rCDI is known to extend the hospitalization length, and to be associated with increased morbidity and mortality rates.

Furthermore, rCDI is often, more than primary infection, associated with life-threatening complications, including pseudomembranous colitis, toxic megacolon, shock, perforation, bloodstream infection (BSI), sepsis, caused by intestinal bacteria or fungi with a mortality rate nearly 50%, and death.

Fecal microbiota transplantation (FMT), defined as the infusion of feces from healthy donors to recipient with disorders associated to dysbiosis, is known to be a highly effective treatment option against CDI. FMT is also more effective than standard treatment with vancomycin and it is recommended by International Guidelines for treating multiple recurrence of CDI.

Despite the increasing body of evidence about the clinical efficacy of FMT for the treatment of rCDI, mechanisms for this clinical efficacy are also unknown.

Metagenomics analysis is known as a good option to examine gut microbiota and to estimate microbial diversity. The aim of this study is to evaluate changes in microbial composition in rCDI patients after FMT, using metagenomics analysis.

DETAILED DESCRIPTION:
Clostridioides diﬃcile infection (CDI) is the most common cause of nosocomial diarrhea, and the most common health care-associated infectious disease in the United States, accounting for 15% of overall infections, nearly 30.000 deaths per year an estimated economic expense of $5 billion/year.

In the last decade, most of the burden related to CDI depends on recurrence CDI (rCDI) (3). rCDI is known to extend the hospitalization length, and to be associated with increased morbidity and mortality rates.

Furthermore, rCDI is often, more than primary infection, associated with life-threatening complications, including pseudomembranous colitis, toxic megacolon, shock, perforation, bloodstream infection (BSI), sepsis, caused by intestinal bacteria or fungi with a mortality rate nearly 50%, and death.

Fecal microbiota transplantation (FMT), defined as the infusion of feces from healthy donors to recipient with disorders associated to dysbiosis, is known to be a highly effective treatment option against CDI. FMT is also more effective than standard treatment with vancomycin and it is recommended by International Guidelines for treating multiple recurrence of CDI.

Despite the increasing body of evidence about the clinical efficacy of FMT for the treatment of rCDI, mechanisms for this clinical efficacy are also unknown.

Metagenomics analysis is known as a good option to examine gut microbiota and to estimate microbial diversity. The aim of this study is to evaluate changes in microbial composition in rCDI patients after FMT, using metagenomics analysis.

The investigators will carry out a single-center observational perspective study. Patients will be recruited among those referred to the gastroenterology unit of the Fondazione Policlinico Universitario "A. Gemelli". Patients with all inclusion criteria and none of the exclusion criteria (detailed in the specific section of this website) will be considered for this study.

Before FMT procedure, demographic data will be collected by the gastrointestinal disease staff.

Moreover, patients will be requested to give stool samples to be collected in a sterile, sealed container and stored at -80°C for metagenomic assessment of gut microbiome and meta-transcriptome assessment by the microbiology staff.

Patients, according to clinical practice, will receive FMT procedure by colonoscopy. Each patient of the study will receive faeces from one single donor without any specific recipient-donor match. The selection of stool donors will be performed by the gastroenterology unit staff following protocols previously recommended by international guidelines and according the new recommendation imposed by the reorganisation of faecal microbiota transplant during the COVID-19 pandemic. All faecal infusates will be manufactured in the microbiology unit of our hospital. Only frozen faeces will be used. Preparation of frozen faeces will follow protocols from international guidelines.

Follow-up visits will be performed by physicians from the gastroenterology unit. All patients will be followed up for 3 months after the end of treatments.

Follow-up visits will be scheduled at week 1, week 2, week 4, and week 12, after the end of treatments. At each visit investigators will collect stool samples for microbiome analysis.

Study Outcomes are detailed in the specific section of this website. For microbiome analysis, statistical differences between group means will be calculated using a two-tailed Wilcoxon-Rank Sum Test, through the R statistical software package (R Core Team, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Recurrent Clostridioides difficile infection
* Age between 18 and 90 years old
* Ability to provide written informed consent
* Ability to be compliant with the scheduled procedures

Exclusion Criteria:

* Another known gastrointestinal infection apart from C. difficile infection

  . Known active gastrointestinal disorders (e.g. infectious gastroenteritis, coeliac disease, inflammatory bowel disease, irritable bowel syndrome, chronic pancreatitis, biliary salt diarrhoea)
* Previous colorectal surgery or cutaneous stoma
* Current or recent (< 6 weeks) therapy with drugs that could possibly alter gut microbiota (e.g. antimicrobials, probiotics)
* Decompensated heart failure or heart disease with ejection fraction lower than 30%
* Severe respiratory insufficiency
* Psychiatric disorders
* Pregnancy or breastfeeding
* Unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent Clostridioides difficile infection, treated with FMT
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Qualitative and quantitative characteristics of recipients' microbiome 30 days after FMT. | 1 months
  The investigators will evaluate the characteristics of recipients' microbiome, assessed by metagenomics analysis, 30 days after FMT compared with baseline.

SECONDARY OUTCOMES:
Qualitative and quantitative characteristics of recipients' microbiome 7,15,90 days after FMT. | 3 months
  The investigators will evaluate the characteristics of recipients' microbiome, assessed by metagenomics analysis, 7,15,90 days after FMT compared with baseline.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 months
  The number of participants with treatment-related adverse events (assessed by CTCAE v4.0) will be recorded throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Ianiro, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to other researchers
Supporting Information: Study Protocol
Time Frame: data will be available after the completion of the study, for 5 years
Access Criteria: Data will be given upon request to the PI

REFERENCES:
- [Background] Miller BA, Chen LF, Sexton DJ, Anderson DJ. Comparison of the burdens of hospital-onset, healthcare facility-associated Clostridium difficile Infection and of healthcare-associated infection due to methicillin-resistant Staphylococcus aureus in community hospitals. Infect Control Hosp Epidemiol. 2011 Apr;32(4):387-90. doi: 10.1086/659156. PMID 21460491
- [Background] Dubberke ER, Olsen MA. Burden of Clostridium difficile on the healthcare system. Clin Infect Dis. 2012 Aug;55 Suppl 2(Suppl 2):S88-92. doi: 10.1093/cid/cis335. PMID 22752870
- [Background] Falcone M, Russo A, Iraci F, Carfagna P, Goldoni P, Vullo V, Venditti M. Risk Factors and Outcomes for Bloodstream Infections Secondary to Clostridium difficile Infection. Antimicrob Agents Chemother. 2015 Oct 19;60(1):252-7. doi: 10.1128/AAC.01927-15. Print 2016 Jan. PMID 26482315
- [Background] Quraishi MN, Widlak M, Bhala N, Moore D, Price M, Sharma N, Iqbal TH. Systematic review with meta-analysis: the efficacy of faecal microbiota transplantation for the treatment of recurrent and refractory Clostridium difficile infection. Aliment Pharmacol Ther. 2017 Sep;46(5):479-493. doi: 10.1111/apt.14201. Epub 2017 Jul 14. PMID 28707337
- [Background] Cammarota G, Masucci L, Ianiro G, Bibbo S, Dinoi G, Costamagna G, Sanguinetti M, Gasbarrini A. Randomised clinical trial: faecal microbiota transplantation by colonoscopy vs. vancomycin for the treatment of recurrent Clostridium difficile infection. Aliment Pharmacol Ther. 2015 May;41(9):835-43. doi: 10.1111/apt.13144. Epub 2015 Mar 1. PMID 25728808
- [Background] Surawicz CM, Brandt LJ, Binion DG, Ananthakrishnan AN, Curry SR, Gilligan PH, McFarland LV, Mellow M, Zuckerbraun BS. Guidelines for diagnosis, treatment, and prevention of Clostridium difficile infections. Am J Gastroenterol. 2013 Apr;108(4):478-98; quiz 499. doi: 10.1038/ajg.2013.4. Epub 2013 Feb 26. PMID 23439232
- [Background] Debast SB, Bauer MP, Kuijper EJ; European Society of Clinical Microbiology and Infectious Diseases. European Society of Clinical Microbiology and Infectious Diseases: update of the treatment guidance document for Clostridium difficile infection. Clin Microbiol Infect. 2014 Mar;20 Suppl 2:1-26. doi: 10.1111/1469-0691.12418. PMID 24118601
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657